CLINICAL TRIAL: NCT04870216
Title: Evaluation of Practices, Knowledge and Expectations of Medical Students for Intimate Protection
Acronym: STUDENT-PROTEC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-004-STUDENT-PROTEC
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Intimate Protections
Keywords: Intimate protections; Medical student
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical student: Medical student aged more than 18, presenting menstrual cycles, and agreeing to participate in the study.
  Interventions: Other: Questionnaire regarding intimate protections habit.

INTERVENTIONS:
Other: Questionnaire regarding intimate protections habit. — Questionnaire regarding intimate protections habit.
  Other Names: Data collection

SUMMARY:
Intimate protections, designed to absorb menstrual flow during menstruation, are classified into two categories: internal intimate protections (tampon, menstrual cup) and external intimate protections (disposable or washable sanitary pads, panty liner, menstrual panty).

Recently, women's expectations have changed with a demand for transparency regarding intimate protection's composition and potential health risks.

The choice and use of a type of intimate protection will depend on multiple factors specific to each woman. The cost of intimate protectioncould influence patient choice, as disposable sanitary pads are often less expensive.

DETAILED DESCRIPTION:
The primary objective is to describe medical students 's intimate protection practices.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Medical student
* Aged more than 18
* Presenting menstrual cycles
* Agreeing to participate in the study

Exclusion Criteria:

- Aged less than 18

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Medical student
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Use of internal intimate protections | Day 0
  Number of patients using tampon or menstrual cup as hygienic protection
Use of external intimate protections | Day 0
  Number of patients using disposable sanitary pads, washable sanitary pads, panty liner or menstrual panty as hygienic protection

CONTACTS AND LOCATIONS:
Overall Officials: Emilie RAIMOND, Principal Investigator — Université de Reims CHampahne-Ardenne - CHU de Reims
Locations (1):
- Université de Reims Champagne-Ardenne, Reims, France